CLINICAL TRIAL: NCT00216424
Title: An Open Label, Phase II Study of Capecitabine (Xeloda) Plus Conformal Radiotherapy for Patients With Locally Advanced, Non-Metastatic Rectosigmoid Carcinoma
Brief Title: Capecitabine (Xeloda) and Radiation for Patients With Rectosigmoid Carcinoma
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: lack of accrual
Sponsor: James A. Haley Veterans Administration Hospital (U.S. Federal Agency)
Collaborators: Hoffmann-La Roche (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XEL372
Record Dates: First submitted 2005-09-21; First posted 2005-09-22 (Estimated); Last update posted 2007-11-12 (Estimated); Status verified 2007-11

CONDITIONS: Colorectal Cancer
Keywords: Colon cancer; Rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Capecitabine

INTERVENTIONS:
Drug: Capecitabine (Xeloda)

SUMMARY:
This study is designed primarily to establish efficacy and estimate resource utilization. The short-term hypothesis is that the dose of capecitabine (825 mg/m2 twice/day 5 days per week) during the course of radiation therapy is efficacious in locally advanced, non-metastatic rectosigmoid carcinoma and will improve resectability. The long-term working hypothesis is that if 3-D CRT is combined with the potentiating and additive effect of capecitabine one hopes to see improved and durable tumor response and survival with acceptable toxicity. In addition, it is expected that the simplicity of using an oral agent (capecitabine) will be associated with reduced cost and resource utilization.

DETAILED DESCRIPTION:
Patients will all receive the combined treatment of 3-D external radiation therapy plus Xeloda®. External Radiation Therapy to the pelvis, lower abdomen and rectal area will be given once a day, five days a week, Monday through Friday, for about five to six weeks using three dimensional techniques.

Xeloda® (oral chemotherapy) is a pill taken by mouth. This medication will be taken during the course of radiation therapy on days that radiation treatments are given. Xeloda pills will be taken twice daily beginning with the first day of radiation therapy treatments and ending on the last day of radiation therapy treatment.

The following tests and procedures are part of regular medical treatment (standard care) for the disease and are also required for this study:

* physical examinations, sometimes including a digital rectal exam
* blood tests including a (blood) pregnancy test will be done before starting treatment if the patient is a woman able to have children.
* urinalysis
* ECG (heart tracing)
* chest X-ray
* ultrasound, which produces pictures of the rectal area using sound waves· CT scan of the pelvis and abdomen

Some people may need surgery, others may require more chemotherapy, and others may require no additional treatment depending on how their tumor responded to the Xeloda® and radiation therapy treatments.

Patients will also be asked to complete two questionnaires about their fatigue, general quality of life, and bowel functioning.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent prior to study-specific screening procedures, with the understanding that the patient has the right to withdraw from the study at any time, without prejudice.
* Age >18 years
* Ambulatory outpatients (if applicable), with Karnofsky performance status of >60
* Histologically or cytologically confirmed locally advanced nonmetastatic T3-4 N0-3 M0 carcinomas of the rectosigmoid.
* Surgical exploration without resection is permissible.
* Protocol Specific Laboratory Values as defined in section 4.2
* Has a negative serum pregnancy test within 7 days prior to start of therapy (female patients of childbearing potential).
* Have concomitant medications been reviewed with patient to address contraindicated medications described in section 7.8 and have precautions been taken as recommended for each drug? Includes Allopurinol, Cimetidine, Sorivudine and Brivudine, Anticoagulants, Phenytoin, and Laxatives.

Exclusion Criteria:

Patients who fulfill any of the following criteria will be excluded:

* Pregnant or lactating woman. Woman of childbearing potential with either a positive or no pregnancy test at baseline. Woman or men of childbearing potential not using a reliable and appropriate contraceptive method. (Postmenopausal woman must have been amenorrheic for at least 12 months to be considered of non-childbearing potential). Patients will agree to continue contraception for 30 days from the date of the last study drug administration
* Life expectancy < 3 months.
* Serious, uncontrolled, concurrent infection(s).
* Prior unanticipated severe reaction to fluoropyrimidine therapy, or known sensitivity to 5-fluorouracil, or known DPD deficiency.
* Completion of previous chemotherapy regimen < four weeks prior to the start of study treatment, or with related toxicities unresolved prior to the start of study treatment.
* Treatment for other carcinomas within the last five years, except cured non-melanoma skin and treated in-situ cervical cancer.
* Participation in any investigational drug study within 4 weeks preceding the start of study treatment.
* Clinically unstable cardiac disease (e.g. congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmias not well controlled with medication) or myocardial infarction within the last 12 months.
* Evidence of metastases or history of uncontrolled seizures, central nervous system disorders or psychiatric disability judged by the investigator to be clinically significant, precluding informed consent, or interfering with compliance of oral drug intake.
* Other serious uncontrolled medical conditions that the investigator feels might compromise study participation.
* Major surgery within 4 weeks of the start of study treatment, without complete recovery (e.g., delayed wound healing).
* Lack of physical integrity of the upper gastrointestinal tract or malabsorption syndrome.
* Known, existing uncontrolled coagulopathy
* Any of the following laboratory values:

  * Abnormal hematologic values (neutrophils < 1.5 x 109/L, platelet count < 100 x 109/L)
  * Impaired renal function (estimated creatinine clearance <30ml/min as calculated with Cockroft-Gault equation.
* Note: In patients with moderate renal impairment (estimated creatinine clearance 30-50 mL/min) at baseline, a dose reduction to 75% of the capecitabine starting dose is recommended.

  * Serum bilirubin > 1.5 x upper normal limit.
  * ALT (SGOT), AST (SGPT) > 2.5 x upper normal limit (or > 5 x upper normal limit in the case of liver metastases).
  * Alkaline phosphatase > 2.5 x upper normal limit (or > 5 x upper normal limit in the case of liver metastases or > 10 x upper normal limit in the case of bone disease)
* Unwillingness to give written informed consent or HIPAA privacy authorization.
* Unwillingness to participate or inability to comply with the protocol requirements for the duration of the study.
* Patient taking a contraindicated medication(s) described in section 6.2.8 (see inclusion criteria #8 for list of agents) and no appropriate substitute agent is available, or patient unable or refuses to take substitute agent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2005-02; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Tumor response and resectability of tumor following treatment with radiation and capecitabine (Xeloda).

CONTACTS AND LOCATIONS:
Overall Officials: Ismail Kazem, MD, Principal Investigator — James A. Haley Veterans Administration Hospital
Locations (1):
- James A. Haley Veterans Administration Hospital, Tampa, Florida, United States